CLINICAL TRIAL: NCT00110253
Title: A Randomized, Double-Blind, Paired, Placebo Controlled Study Evaluating the Duration of Anesthetic Effect Produced by the S-Caine™ Peel (Lidocaine 7% and Tetracaine 7% Cream) When Applied for 30 and 60 Minutes
Brief Title: Duration of Skin Numbing Effect Created by the S-Caine™ Peel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCP-44-05
Record Dates: First submitted 2005-05-04; First posted 2005-05-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-Caine Peel (Experimental)
  Interventions: Drug: S-Caine™ Peel (lidocaine and tetracaine cream 7%/7%)

INTERVENTIONS:
Drug: S-Caine™ Peel (lidocaine and tetracaine cream 7%/7%) — S-Caine Peel is composed of a 1:1 eutectic mixture of 7% lidocaine, and 7% tetracaine, which was applied topically. The S Caine Peel was applied at approximately 1 mm in thickness and remained on the treatment area for 30 or 60 minutes
  Other Names: Pliaglis

SUMMARY:
S-Caine™ Peel (lidocaine 7% and tetracaine 7% cream) is a new skin numbing cream made of lidocaine and tetracaine. The purpose of this study is to evaluate and measure the length of time the S-Caine Peel numbs the skin, when applied for 30 and 60 minutes.

DETAILED DESCRIPTION:
This was a single center, randomized, double-blind, placebo controlled, paired study that evaluated the duration of anesthetic effect produced by S-Caine Peel when applied for 30 or 60 minutes in 40 adult volunteers. A pinprick test was used to determine duration of anesthetic effect.

At the procedure visit, subjects were to be assigned the lowest available sequential subject number. Treatment was randomized according to a computer-generated randomization schedule provided by the sponsor. The randomization to application time of 30 or 60 minutes was to be 1:1 and un-blinded. The randomization of study drug to treatment area (concurrent applications of either S Caine Peel applied to the anterior surface of the right thigh with placebo applied to the anterior surface of the left thigh, or placebo applied to the anterior surface of the right thigh and S-Caine Peel applied to the anterior surface of the left thigh) was 1:1 and double-blind. Instructions for implementing the randomization (ie, the correct application time and treatment area) appeared on the study drug labels assigned to each subject number.

Subjects were administered both S-Caine Peel and placebo on separate thighs for either 30 or 60 minutes. The study drugs were applied concurrently to the anterior surfaces of the right and left thigh (one application per thigh, with study drug applied to the right thigh first, followed immediately by application of the alternate study drug to the left thigh). Each study drug was dispensed to cover a 200 cm² treatment area with a uniform thickness of approximately 1 mm

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older.
* Meet pinprick test requirements.

Exclusion Criteria:

* Subject is pregnant or breastfeeding.
* Subject has participated in a clinical trial of an unapproved drug within the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Duration of anesthetic effect | first time after onset when the number of painful pinpricks was 3 or more for 2 consecutive time points
  The duration of anesthesia was defined as the difference between the onset and end of anesthesia. If there was no onset of anesthesia, the duration was defined as zero. Onset of anesthesia was defined as the first time that the number of painful pinpricks was 2 or less (out of 5) for 2 consecutive time points. For subjects/treatments with onset of anesthesia, the end of anesthesia was defined as the first time after onset when the number of painful pinpricks was 3 or more for 2 consecutive time points

SECONDARY OUTCOMES:
Number of participants with adverse events | 72 hours
  To monitor the nature and frequency of adverse events (AEs) associated with the application of S-Caine Peel

CONTACTS AND LOCATIONS:
Overall Officials: William Garland, MD, Principal Investigator — Radiant Research San Diego
Locations (1):
- Radiant Research, San Diego, California, United States